CLINICAL TRIAL: NCT04456413
Title: Phase II Randomized Study of Convalescent Plasma From Recovered COVID-19 Donors Collected by Plasmapheresis as Treatment for Subjects With Early COVID-19 Infection
Brief Title: Convalescent Plasma as Treatment for Subjects With Early COVID-19 Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Hackensack Meridian Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020-0542
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: Coronavirus; Covid19; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma (Experimental): Fresh or frozen plasma will be infused one time to patients
  Interventions: Biological: Convalescent Plasma
- Best Supportive Care (Active Comparator): Patients will receive best supportive care. Patients randomized to best supportive care may receive plasma should they require hospitalization for progression of COVID-19 disease.
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Biological: Convalescent Plasma — Fresh or frozen plasma will be infused one time to hospitalized patients with COVID-19 infection
  Arms: Convalescent Plasma
Other: Best Supportive Care — Patients will receive best supportive care. Patients randomized to this arm may receive plasma should they require hospitalization for progression of COVID-19 disease.
  Arms: Best Supportive Care

SUMMARY:
* This is a phase II randomized study of convalescent plasma for the treatment of non-immune individuals with COVID-19 infection at high risk of complications.
* Subjects will be considered as having completed the study after 2 months (+/- 5) days, unless consent withdrawal or death occurs first.
* Subjects will be randomized to receiving convalescent plasma or best supportive care.
* Patients randomized to best supportive care may receive plasma should they require hospitalization for progression of COVID-19 disease.
* The final analysis will be conducted once the last subject completes the 2-month visit or withdraws from the study.

DETAILED DESCRIPTION:
Overall study design

* This is a phase II randomized study of convalescent plasma for the treatment of non-immune individuals with COVID-19 infection at high risk of complications.
* Subjects will be considered as having completed the study after 2 months (+/- 5) days, unless consent withdrawal or death occurs first.
* Subjects will be randomized to receiving convalescent plasma or best supportive care.
* Patients randomized to best supportive care may receive plasma should they require hospitalization for progression of COVID-19 disease.
* The final analysis will be conducted once the last subject completes the 2-month visit or withdraws from the study.

A total of 306 subjects will be recruited, 153 for each arm. If a patient in the best supportive care arm requires hospitalization, the patient will be eligible to receive convalescent plasma if requested and/or deemed medically appropriate by the admitting physician.

Overall study duration

* The study begins when the first subject (donor or recipient) signs the informed consent. The study will end once the last enrolled subject completes the study (likely a recipient).
* The expected duration of the study is approximately 12 months.

ELIGIBILITY:
Donor Eligibility Criteria:

* Age 18-60
* A history of a positive nasopharyngeal swab for COVID-19 or a history of positive antibody titer test.
* At least 14 days from resolution of COVID-19-associated symptoms including fevers.
* A negative nasopharyngeal swab (or similar test) for COVID-19
* anti-SARS-CoV2 titers >1:500
* Adequate venous access for apheresis
* Meets donor eligibility criteria in accordance to Hackensack University Medical Center (HUMC) Collection Facility at the John Theurer Cancer Center (JTCC) if collecting at the JTCC, and all regulatory agencies as describes in SOP 800 01.
* Required testing of the donor and product must be performed in accordance to FDA regulations (21 CFR 610.40), and the donation must be found suitable (21 CFR 630.30)

Recipient Eligibility Criteria:

* Patient age >30 years old, newly diagnosed with a COVID-19 infection with onset of first symptoms < 96 hours.
* And least one other high-risk feature:

  1. Age > 65
  2. BMI 30 or above
  3. Hypertension, defined as SBP above 140 or DBP above 90, or requiring medication for control.
  4. Coronary artery disease (history, not ECG changes only)
  5. Congestive heart failure
  6. Peripheral vascular disease (includes aortic aneurysm >= 6 cm)
  7. Cerebrovascular disease (history of CVA or TIA)
  8. Dementia
  9. Chronic pulmonary disease
  10. Liver disease (such as portal hypertension, chronic hepatitis)
  11. Diabetes (excludes diet-controlled alone)
  12. Moderate or severe renal disease defined as having a GFR < 60 mL/min
  13. Cancer (exclude if > 5 year in remission)
  14. AIDS (not just HIV positive)

Recipient exclusion criteria:

* History of severe transfusion reaction to plasma products
* Need for oxygen supplementation
* Positive test for COVID-19 antibodies
* Chemotherapy-induced neutropenia (ANC < 0.5 x 103/mcL)
* Immunosuppressive medications except for prednisone (or steroid equivalent) > 10 mg daily.
* Performance status < 50 by KPS
* Pneumonia by radiographic evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Donato, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Casadevall A, Scharff MD. Return to the past: the case for antibody-based therapies in infectious diseases. Clin Infect Dis. 1995 Jul;21(1):150-61. doi: 10.1093/clinids/21.1.150. PMID 7578724
- [Background] Casadevall A, Pirofski LA. Antibody-mediated regulation of cellular immunity and the inflammatory response. Trends Immunol. 2003 Sep;24(9):474-8. doi: 10.1016/s1471-4906(03)00228-x. No abstract available. PMID 12967670
- [Background] Casadevall A, Dadachova E, Pirofski LA. Passive antibody therapy for infectious diseases. Nat Rev Microbiol. 2004 Sep;2(9):695-703. doi: 10.1038/nrmicro974. PMID 15372080
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Zhang JS, Chen JT, Liu YX, Zhang ZS, Gao H, Liu Y, Wang X, Ning Y, Liu YF, Gao Q, Xu JG, Qin C, Dong XP, Yin WD. A serological survey on neutralizing antibody titer of SARS convalescent sera. J Med Virol. 2005 Oct;77(2):147-50. doi: 10.1002/jmv.20431. PMID 16121363
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Yeh KM, Chiueh TS, Siu LK, Lin JC, Chan PK, Peng MY, Wan HL, Chen JH, Hu BS, Perng CL, Lu JJ, Chang FY. Experience of using convalescent plasma for severe acute respiratory syndrome among healthcare workers in a Taiwan hospital. J Antimicrob Chemother. 2005 Nov;56(5):919-22. doi: 10.1093/jac/dki346. Epub 2005 Sep 23. PMID 16183666
- [Background] Ko JH, Seok H, Cho SY, Ha YE, Baek JY, Kim SH, Kim YJ, Park JK, Chung CR, Kang ES, Cho D, Muller MA, Drosten C, Kang CI, Chung DR, Song JH, Peck KR. Challenges of convalescent plasma infusion therapy in Middle East respiratory coronavirus infection: a single centre experience. Antivir Ther. 2018;23(7):617-622. doi: 10.3851/IMP3243. Epub 2018 Jun 20. PMID 29923831
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] Gunn BM, Yu WH, Karim MM, Brannan JM, Herbert AS, Wec AZ, Halfmann PJ, Fusco ML, Schendel SL, Gangavarapu K, Krause T, Qiu X, He S, Das J, Suscovich TJ, Lai J, Chandran K, Zeitlin L, Crowe JE Jr, Lauffenburger D, Kawaoka Y, Kobinger GP, Andersen KG, Dye JM, Saphire EO, Alter G. A Role for Fc Function in Therapeutic Monoclonal Antibody-Mediated Protection against Ebola Virus. Cell Host Microbe. 2018 Aug 8;24(2):221-233.e5. doi: 10.1016/j.chom.2018.07.009. PMID 30092199
- [Background] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Crowe JE Jr, Firestone CY, Murphy BR. Passively acquired antibodies suppress humoral but not cell-mediated immunity in mice immunized with live attenuated respiratory syncytial virus vaccines. J Immunol. 2001 Oct 1;167(7):3910-8. doi: 10.4049/jimmunol.167.7.3910. PMID 11564809
- [Background] Tan M, Xiong X. Continuous and group sequential conditional probability ratio tests for phase II clinical trials. Stat Med. 1996 Oct 15;15(19):2037-51. doi: 10.1002/(SICI)1097-0258(19961015)15:193.0.CO;2-Z. PMID 8896138
- [Background] Tan MT, Xiong X. A flexible multi-stage design for phase II oncology trials. Pharm Stat. 2011 Jul-Aug;10(4):369-73. doi: 10.1002/pst.478. Epub 2010 Dec 8. PMID 22328328
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Treanor JJ, Hayden FG, Vrooman PS, Barbarash R, Bettis R, Riff D, Singh S, Kinnersley N, Ward P, Mills RG. Efficacy and safety of the oral neuraminidase inhibitor oseltamivir in treating acute influenza: a randomized controlled trial. US Oral Neuraminidase Study Group. JAMA. 2000 Feb 23;283(8):1016-24. doi: 10.1001/jama.283.8.1016. PMID 10697061
- [Background] Austin SR, Wong YN, Uzzo RG, Beck JR, Egleston BL. Why Summary Comorbidity Measures Such As the Charlson Comorbidity Index and Elixhauser Score Work. Med Care. 2015 Sep;53(9):e65-72. doi: 10.1097/MLR.0b013e318297429c. PMID 23703645
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Convalescent Plasma | Best Supportive Care
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convalescent Plasma | Best Supportive Care | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Hospitalization Rate
Description: The hospitalization rate will be summarized by frequency (%) and compared between the Treatment and Control arms by Mantel-Haenszel test.
Time Frame: 10 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Best Supportive Care
Number analyzed (Participants) | 10 | 11
Participants | 1 | 3

2. Secondary Outcome: Time to Symptoms Resolution
Description: The time to symptoms resolution is defined as the time in days from therapies initiation to the first documented symptoms resolution as assessed by a local site. Patients whose symptoms are not resolved, or result in death, or lost follow-up on the designed follow-up date, will be censored on that date.
Time Frame: 2 Months
Population: Due to a lack of funding and early termination of the trial, these data were not collected.
Arm/Group | Convalescent Plasma | Best Supportive Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival Rate
Description: Overall survival (OS) will be defined as Rate of death
Time Frame: 2 Months
Measure: Number; unit: Patient Deaths
Arm/Group | Convalescent Plasma | Best Supportive Care
Number analyzed (Participants) | 10 | 11
Patient Deaths | 0 | 0

4. Secondary Outcome: Rate of Virologic Clearance by Nasopharyngeal Swab at 2 Weeks
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Best Supportive Care
Number analyzed (Participants) | 10 | 9
Participants | 6 | 6

5. Secondary Outcome: Rate of Nasopharyngeal Swab Positivity in Donors
Time Frame: 2 Months
Population: Due to a lack of funding and early termination of the trial, these data were not collected.
Arm/Group | Convalescent Plasma | Best Supportive Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Rate of Donor Titers Level
Description: Rate of Donor Titer Levels >1:1000
Time Frame: 2 Months
Measure: Count of Participants; unit: Participants
Groups:
- Convalescent Plasma Donors: Convalescent Plasma Donors
Arm/Group | Convalescent Plasma Donors
Number analyzed (Participants) | 69
Participants | 55

7. Secondary Outcome: Impact of Donor Titers Level on Efficacy
Time Frame: 2 Months
Population: Due to a lack of funding and early termination of the trial, these data were not collected.
Arm/Group | Convalescent Plasma | Best Supportive Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patients' Anti-SARS-CoV2 Titer Assessment Pre-infusion for the Treatment Group, at 2 Weeks , 4 Weeks and 2 Months.
Time Frame: Prior to treatment, 2 Weeks, 4 Weeks, and 2 Months
Population: Due to a lack of funding and early termination of the trial, these data were not collected.
Arm/Group | Convalescent Plasma | Best Supportive Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Rate of Virologic Clearance by Nasopharyngeal Swab at 4 Weeks
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Best Supportive Care
Number analyzed (Participants) | 6 | 4
Participants | 5 | 2

10. Other Pre Specified Outcome: Plasma Product's Cytokine Level Assessment
Description: Univariate test will be performed in terms of identifying the association between exploratory objective and the hospitalization rate, Mantel-Haenszel test for categorical variables, and t-test or its non-parametric version for the continuous variables based on the normalized of the data.
Time Frame: Day 0
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Plasma Product's Mannose-binding Lectin (MBL) Level Assessment
Time Frame: Day 0
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Plasma Product's Procalcitonin (PCT) Level Assessment
Time Frame: Day 0
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Plasma Product's C-reactive Protein (CRP) Level Assessment
Time Frame: Day 0
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Plasma Product's Human Neutrophil Lipocalin (HNL) Level Assessment
Time Frame: Day 0
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Plasma Product's Annexin V Level Assessment
Time Frame: Day 0
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Plasma Product's Surfactant Protein D (SP-D) Level Assessment
Time Frame: Day 0
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Plasma Product's microRNA Level Assessment
Time Frame: Day 0
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Plasma Product's Immunoglobulin Level Assessment
Time Frame: Day 0
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Patients' Cytokines Levels Assessment at +2 and +4 Weeks Post Randomization
Time Frame: 2 Weeks and 4 Weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Patients' Chemokines Levels Assessment at +2 and +4 Weeks Post Randomization
Time Frame: 2 Weeks and 4 Weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Rates of Adverse Events Associated With Convalescent Plasma Infusion.
Description: Safety assessment will be performed on infusion day for the Treatment group (immediately post infusion), and for all patients on randomization day +3 and +7 days (by telephone, closest business day is acceptable), +2 weeks (+/- 3 days), +4 weeks (+/- 3 days).
Time Frame: Day 3 and 7, Weeks 2 and 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Arm/Group | Convalescent Plasma | Best Supportive Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/11
Other Adverse Events (participants affected / at risk) | 1/10 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Convalescent Plasma (N=10) | Best Supportive Care (N=11)
Worsening Covid Symptoms (Infections and infestations) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Convalescent Plasma (N=10) | Best Supportive Care (N=11)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The convalescent plasma technology has been replaced by antivirals and monoclonal antibodies. Therefore, the study was not able to accrue successfully and was subsequently terminated. All available data (due to the lack of a formal analysis) is reported here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT04456413/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT04456413/ICF_000.pdf